CLINICAL TRIAL: NCT05780333
Title: Effect of Erector Spinae Plane Block and Transversus Abdominis Plane Block on Quality of Recovery and Postoperative Pain After Laparoscopic Hysterectomy; Randomized, Double-blinded Clinical Trial
Brief Title: Effect of Different Plane Blocks on Quality of Recovery and Postoperative Pain After Laparoscopic Hysterectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mentese State Hospital (Other Government)
Responsible Party: Principal Investigator, Pelin Dilsiz Eker, MD., specialist, Mentese State Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/12
Record Dates: First submitted 2023-03-04; First posted 2023-03-22 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Post Operative Pain
Keywords: tap block; esp block; postoperative pain; recovery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is a double blind, randomized control clinical trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple (Participant, Care Provider, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tap block (Other): Tap block is one of the frequently used field blocks for analgesia management of abdominal surgery.
  At the end of surgery and general anesthesia, transversus abdominis fascial plane will be detected with using lineer usg probe. With in-plane tecnique after placement of the needle in the transversus abdominis fascial plane, and careful aspiration to exclude vascular puncture, a test dose of 1 mL will be injected to determine resistance to flow, and confirm needle tip placement within the fascial plane. After this, 20 ml local anaestetic mixture will be injected through the needle. The TAP block will be then performed on the opposite side using an identical technique.
  Interventions: Procedure: TAP block
- esp block (Active Comparator): The effectiveness of esp block is also evaluated in abdominal surgery after spinal surgery, thoracic and cardiovascular surgery.
  At the end of surgery and general anesthesia, in the lateral decubitus position, the linear probe will be placed approximately 3 cm lateral to the T10 spinous process, in the parasagittal plane. With the in-plane technique, when the block needle rests on the transverse process (approximately 3cm in depth), the erector spina plan will be confirmed with a 0.5-1 mL 0.9% NaCl test dose. 20 ml of local anesthetic mixture will be applied to the confirmed area. The procedure will be applied bilaterally.
  Interventions: Procedure: ESP block

INTERVENTIONS:
Procedure: TAP block — Bilateral tap block with 20 ml of mixture 2:1:1 (0.5% bupivacaine: 0.9%NaCl: 2% lidocain) for each
  Arms: tap block
Procedure: ESP block — Bilateral esp block with 20 ml of mixture 2:1:1 (0.5% bupivacaine: 0.9%NaCl: 2% lidocain) for each
  Arms: esp block

SUMMARY:
The goal of this clinical trial is to evaluate in effect of tap block and esp block on quality of recovery and postoperative pain after laparoscopic hysterectomy. The main question it aims to answer are: Are these two plane blocks used superior to each other? Participants;

* will fill out the preoperative questionnaire
* will fill out the postoperative questionnaire
* will report their pain status according to the NRS score

DETAILED DESCRIPTION:
Standard management of acute pain after surgery consists mainly of systemic opioid narcotics and nonsteroidal anti-inflammatory drugs (NSAIDs). Generally, opiates and NSAIDs are not completely effective at managing pain, and they carry significant risk of addiction and overdose, particularly with prolonged or increased dosing. The concept of multimodal or ''balanced'' analgesia is rapidly becoming the 'standard of care' for preventing post-operative pain. It consists of the use of combinations of analgesics of different classes with different sites of action in an attempt to provide superior pain relief with reduced analgesic related side effects. Local anesthetic injection to block specific nerves has been widely recognized as a useful adjunct in a multimodal approach to postoperative pain management.

Erector Spinae Plane (ESP) block is a recently described plane block designed to block the dorsal and ventral rami of the spinal nerves. And this block provides visceral and somatic pain block.

Transversus Abdominis plane (TAP) block involves the injection of LA between the transversus abdominis (TA) and internal oblique (IO) muscles.This interfascial plane contains the intercostal, subcostal, iliohypogastric, and ilioinguinal nerves. These nerves give sensation to the anterior and lateral abdominal wall as well as the parietal peritoneum, providing only somatic and not visceral analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Female patients who will undergo hysterectomy under elective conditions
* 18- 65 years
* ASA I-II patients

Exclusion Criteria:

* Refusal during registration, request to be excluded from the study, failure to give informed consent
* Under 18 years old and upper 65 years old
* ASA III-IV patients
* Chronic opioid use
* Presence of infection at the injection site
* Renal failure / Liver failure
* Bupivacaine sensitivity
* Use of anticoagulants
* BMI < 18,5 , BMI >35

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — It will be planned for female gender as patients who have undergone hysterectomy will be selected.
Enrollment: 60 (Estimated)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery 40 Questionnaire | 24 hours after surgery.
  The global Quality of Recovery-40 aggregate score is a scale from (1 to 5, where: 1 = very poor and 5 = excellent)

SECONDARY OUTCOMES:
Postoperative pain | 24 hours after surgery.
  is a numerical rating scale from (1 to 10, where: 1 is the mildest and 10 the worst possible)

OTHER OUTCOMES:
using salvage opiod | 24 hours after surgery.
  Additional opioid use for nrs score of 4 and above

CONTACTS AND LOCATIONS:
Overall Officials: pelin dilsiz eker, MD, Principal Investigator — Mentese State Hospital; Ismail Gökbel, MD, Study Chair — Mentese State Hospital; Sinem Sari Ozturk, MD, Study Director — Aydin Adnan Menderes University, Department of anesthesiology and reanimation
Locations (1):
- Pelin Dilsiz Eker, Muğla, Menteşe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yap JY, Bhat M, McMullen W, Ragupathy K. Novel use of laparoscopic-guided TAP block in total laparoscopic hysterectomy. J Obstet Gynaecol. 2018 Jul;38(5):736. doi: 10.1080/01443615.2018.1444402. PMID 29944049
- [Result] Rosato C, Santonastaso DP, de Chiara A, Viola L, Russo E, Piccioni FG, Agnoletti V. Erector spinae plane block for pain management in laparoscopic hysterectomy and bilateral oophorectomy. J Clin Anesth. 2021 Jun;70:110184. doi: 10.1016/j.jclinane.2021.110184. Epub 2021 Feb 6. No abstract available. PMID 33561705
- [Result] Yagi K, Adachi K, Tanaka E, Toda A, Miyoshi Y, Funada R, Yamamoto Y. The Role of Preoperative and Postoperative Transversus Abdominis Plane and Rectus Sheath Block in Patients Undergoing Total Laparoscopic Hysterectomy. J Perianesth Nurs. 2020 Oct;35(5):491-495. doi: 10.1016/j.jopan.2020.02.014. Epub 2020 Jun 18. PMID 32565029
- See also: Erector spinae plane block for pain management in laparoscopic hysterectomy and bilateral oophorectomy — https://pubmed.ncbi.nlm.nih.gov/33561705/
- See also: The Role of Preoperative and Postoperative Transversus Abdominis Plane and Rectus Sheath Block in Patients Undergoing Total Laparoscopic Hysterectomy — https://pubmed.ncbi.nlm.nih.gov/32565029/
- See also: Novel use of laparoscopic-guided TAP block in total laparoscopic hysterectomy — https://pubmed.ncbi.nlm.nih.gov/29944049/

DOCUMENTS (2):
  • Informed Consent Form: Informed Consent Form / ESP arm (2023-01-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT05780333/ICF_000.pdf
  • Informed Consent Form: Informed Consent Form / TAP arm (2023-01-21): https://cdn.clinicaltrials.gov/large-docs/33/NCT05780333/ICF_001.pdf